CLINICAL TRIAL: NCT05226182
Title: Visualisation of a Digital Care Pathway in Limburg, in Context of Digital Care Support as a Stepping Stone for Flanders.
Brief Title: Visualisation of a Digital Care Pathway.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jessa Hospital (Other)
Collaborators: Wit-Gele Kruis Limburg (Unknown); KLAV (Unknown); Ferm Thuiszorg (Unknown); I-mens (Unknown); Vlaams Patiëntenplatform (Unknown); Wit-Gele Kruis Vlaanderen (Unknown); POM Limburg (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021/036
Record Dates: First submitted 2021-10-27; First posted 2022-02-07 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes; Multidisciplinary Communication; Empowerment; Patient Empowerment; Patient Acceptance of Health Care
Keywords: digital; care; pathway; type 2; Diabetes; visualization; E-health; pilot study; visualisation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Empowerment; Patient Participation; Patient Acceptance of Health Care; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The patient population in this pilot study consists of two cohorts. All inclusions start from the GP, based on well-defined inclusion criteria. The reason for working with two parallel cohorts is based on the premise that different patient characteristics will confound the results and provide a distorted conclusion if not separated. One group is anticipated to consist of patients capable of using the application independently, while the other group is expected to have patients that will likely be more dependent on others for help with digital applications. This discrepancy could impact the usability and evaluation of the application.
  Literature shows that in similar pilot studies numbers of participants can vary a lot. Taking into regard the inclusion criteria, labor intensity and limited resources of this study investigators aim to include 15-30 patients for cohort 1 and 5-15 patients for cohort 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients (Experimental): Implementation and visualisation of digital care path. Pre measurement: questionnaire quantifying patient involvement and experience on a 5-p Likert scale.
  Post measurement: questionnaire quantifying patient involvement and experience on a 5-p Likert scale, questionnaire quantifying usability of the tool and in-depth interview.
  Interventions: Other: visualisation of a digital care path
- healthcare professionals (Experimental): Implementation and visualisation of digital care path. Pre measurement: questionnaire quantifying communication needs and experiences on a 5-p Likert scale.
  Post measurement: questionnaire quantifying communication needs and experiences on a 5-p Likert scale, questionnaire quantifying usability of the tool and in-depth interview.
  Interventions: Other: visualisation of a digital care path

INTERVENTIONS:
Other: visualisation of a digital care path — The implementation and visualisation of a digital care path, specifically designed for patients with type 2 diabetes and their care team. The digital care path wil include: 1) a timeline with appointments, messages and questionnaires 2) Diabetes related articles 3) a page for monitoring clinical parameters and goals 4) a section displaying information on their care team and personal health records. The aim of this intervention is to evaluate whether providing a central platform for all data will increase patient empowerment and involvement. Secondly it will also evaluate whether the communication between healthcare professionals improves when selected data is readily available for the entire care team.

SUMMARY:
As part of the EFRO (Europees Fonds Regionale Ontwikkeling) 1302 project "Digital Care Support in Practice with Limburg as a Stepping Stone for Flanders", this study aims to evaluate the concept and added value of visualising a personal digital care pathway for patients with type 2 diabetes. Firstly, this chronological visualisation of data strives to improve patient experience and empowerment by offering educational articles and personal medical data relevant to their care path in one place. This way, patients will have more insight in the pathogenesis, treatments, complications and goals, allowing the patients to optimize their selfcare and become confident in dealing with their chronic condition. From time to time, patients will also be asked to complete questionnaires concerning their experiences (PREM) to aid healthcare professionals in personalizing treatment goals. Secondly, the healthcare providers and caregivers surrounding the patient will also have access to the same data, allowing for a more personal approach as well as means to communicate with other members of the care team.

DETAILED DESCRIPTION:
Good quality of care requires a multidisciplinary approach, especially with chronic illnesses. Therefore, all members of the care team should be adequately informed and communicate well with each other. Additionally, patients should have a key role in their treatment plan. To successfully optimize self care, patients have to be well-informed about pathogenesis, treatments and complications so that expectations are realistic and attainable goals can be set. Currently, access to this relevant data is fragmented and often unavailable.

The newly developed application creates a central platform where all relevant data, educational material, medication scheme... are available for both the patient and healthcare professionals. The targeted study population are patients with type 2 diabetes who will be recruited by their general practitioner (GP) over a period of 3 months. When patients are interested in partaking, they will be contacted by a healthcare professional who will function as a Single Point of Contact (SPOC) for the patient during the entirety of the study with a maximum duration of 6 months. The SPOC helps with the start up of the application, collects administrative data and contacts the participants at regular intervals to help with difficulties in using the application. Furthermore, the SPOC will administer a questionnaire determining patient involvement and experience at the start and end of the study, as well as conduct an in-depth interview when the study is completed. Throughout the study, other questionnaires will be digitally available for the patient as part of the care path. These patient reported outcome and experience measures (PROM/PREM) will support healthcare professionals in providing a more integral care.

Consequently, involved healthcare professionals will also be contacted, informed and asked to complete a questionnaire once healthcare professionals agree to participate in the study. This questionnaire will focus on the information and communication needs between members of the care team and will also be repeated at the end, followed by an in-depth interview.

ELIGIBILITY:
Inclusion Criteria for cohort 1 and 2:

* patients with type 2 diabetes (voortraject and zorgtraject)
* independent and mentally competent
* digitally literate and in possession of an email address
* mastered the Dutch language
* able to visit the GP (no house calls)

Additional inclusion criteria for cohort 2 :

* presence of a home nurse in the context of the Diabetes care
* presence of a home care service

Exclusion Criteria:

* patients type 2 Diabetes enrolled in the Diabetes convention
* pregnant patients
* illiterate people
* patients living in a residential care center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in patient empowerment and involvement | For a minimum of 12 weeks
  Primary outcome measures will be determined with the aid of a questionnaire scoring answers on a 5p-Likert scale. Due to limited availability of validated questionnaires in Dutch, a custom set of questions was generated. Starting from validated English questionnaires on each topic, the Delphi method was used to reach consensus in selecting the final questions.
  At the end of the study, an in-depth interview will take place with a predefined topic list.
Change in care team communication and sharing of data | For a minimum of 12 weeks
  Primary outcome measures will be determined with the aid of a questionnaire scoring answers on a 5p-Likert scale. Due to limited availability of validated questionnaires in Dutch, a custom set of questions was generated. Starting from validated English questionnaires on each topic, the Delphi method was used to reach consensus in selecting the final questions.
  At the end of the study, an in-depth interview will take place with a predefined topic list.
Usability and acceptance of the application in patients and healthcare professionals | For a minimum of 12 weeks
  Primary outcome measures will be determined with the aid of a questionnaire scoring answers on a 5p-Likert scale. Due to limited availability of validated questionnaires in Dutch, a custom set of questions was generated. Starting from validated English questionnaires on each topic, the Delphi method was used to reach consensus in selecting the final questions.
  At the end of the study, an in-depth interview will take place with a predefined topic list.

SECONDARY OUTCOMES:
User characteristics of the application. | for a minimum of 12 weeks
  Data will be collected from logs, available in the back office of the application
Possible change,impact on personal clinical parameters: HbA1c | for a minimum of 12 weeks
  HbA1c will be expressed in %
Possible change,impact on personal clinical parameters: blood pressure | For a minimum of 12 weeks
  Both systolic and diastolic blood pressure will be measured, expressed in mmHg.
Possible change,impact on personal clinical parameters: glycemia | For a minimum of 12 weeks
  Glycemia will be expressed in mg/dl.
Possible change,impact on personal clinical parameters: girth | For a minimum of 12 weeks
  Girth will be expressed in cm.
Possible change,impact on personal clinical parameters: bodyweight | For a minimum of 12 weeks
  Weight will be expressed in kg.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Breysem, Dr, Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No